CLINICAL TRIAL: NCT04696718
Title: Determination of the Biological Activity of Serum From Patients With Rheumatoid Arthritis After Consumption of Three Different Probiotics Strains (Lactobacillus Salivarius, Rhamnosus, Bifidobacterium Lactis)
Brief Title: Determination of the Biological Activity of Serum From Patients
Acronym: nutricell3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Adeline BLOT (Other)
Collaborators: Centre Hospitalier Emile Roux (Other); Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government)
Responsible Party: Sponsor-Investigator, Adeline BLOT, Clinical Research Associate, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Organization: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-A00303-52
Record Dates: First submitted 2020-12-07; First posted 2021-01-06 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Women; Rheumatoid Arthritis
Keywords: rheumatoid arthritis; probiotics
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Crossover Assignment patient may receive 3 products in 3 interventions sequentially during the protocol
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traitement 1 (Experimental): Lactobacillus salivarius
  Interventions: Dietary Supplement: daily supplementation
- Traitement 2 (Experimental): Lactobacillus Rhamnosus GG
  Interventions: Dietary Supplement: daily supplementation
- Traitement 3 (Experimental): Bifidobacterium lactis
  Interventions: Dietary Supplement: daily supplementation

INTERVENTIONS:
Dietary Supplement: daily supplementation — the patients will consume 1 pill of probiotic each day for 28 days per treatments each treatment is separated by a wash out period of 21 days

SUMMARY:
The main objective of the study is to determine the influence of patient sera before and after probiotic intervention on the behavior of bone cells (osteoblasts and osteoclasts).

The secondary objectives are to assess the activity of bone cells and the course of rheumatoid arthritis before and after the consomption of probiotics.

DETAILED DESCRIPTION:
The written consent of the subjects will be obtained after full information of the aims, nature and possible risks of the study.

Before inclusion, subjects will undergo a medical check-up including an interview on personal and family history and drug treatments taken as well as a standard medical examination including weight, height and blood pressure measurement. . Their compliance with the inclusion / exclusion criteria will be verified during this review. An interview with personnel involved in the research (a dietician / study Research clinic assistant, etc.) will also be carried out as well as a biological selection assessment.

As part of this study, the subjects will come a total of 7 times to the Emile ROUX hospital in Le Puy en Velay.

The probiotic treatment will begin between 1 and 3 weeks after the inclusion visit. The volunteers / patients recruited will have a volume of blood sampled and a stool collected before the start of the probiotic treatment (T = 0) and at the end of the treatment (T = 4 weeks). The study consists of three periods of probiotic treatment of 4 weeks each interspersed with a wash-out period of 3 weeks in accordance with the recovery period necessary between two blood samples.

The sera thus obtained will then be analyzed to determine their biological activity with regard to the induction of changes in the behavior of bone cell models: osteoformin cells (osteoblasts) and osteo-resorbent cells (osteoclasts).

ELIGIBILITY:
Inclusion Criteria:

Women

* 30-75 years
* Non-menopausal or menopausal for more than 2 years because the tissue osteoarticular is under the influence of steroid hormones. Peri-menopause is accompanied by strong hormonal variations.
* With rheumatoid arthritis (DAS28 threshold specified below)
* Clinical arthritis score ≥ 2.6 (DAS28). Pathology needs to be characterized even if the score remains low
* Person with good venous condition

Exclusion Criteria:

Vaccination in the last two months

* Alcohol abuse with regard to WHO standards
* Smoking (>5 cigarettes/day)

  -> 5 hours of intense sport per week
* Food allergy and others
* Antibiotic treatment in the month preceding inclusion
* Persons under guardianship, curators, deprived of liberties, safeguard of justice
* Refusal to sign the information and consent form

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — higher prevalency of RA in women
Enrollment: 20 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2022-12-22 (Estimated); Study Completion 2023-12-28 (Estimated)

PRIMARY OUTCOMES:
Change of biological activity of serum between day 0 to day 28 | Day 0 and Day 28
  Ex vivo quantification of the formation of osteoclast multi-nucleated cells following culture in the presence of metabolites from the serum of patients between day 0 and day 28

SECONDARY OUTCOMES:
Change of Disease Activity Score (DAS28) day 0 to day 28 | Day 0 and Day 28
  The Disease Activity Score (DAS) is a combined index to measure the disease activity in patients with rheumatoid arthritis (RA).
  Evaluation of a patient's response to treatment can be made much easier and more objective using the DAS28. (Twenty-eight tender and swollen joint scores include the same joints: shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints and the knees.) Simply assess the number of swollen and tender joints and measure the ESR. The DAS will provide you with a number between 0 and 10, indicating the activity rate of the rheumatoid arthritis is at that particular moment.

CONTACTS AND LOCATIONS:
Overall Officials: benjamin castagne, MD, Principal Investigator — Centre Hospitalier Emile Roux
Locations (1):
- Centre Hospitalier Emile Roux, Le Puy-en-Velay, France

IPD SHARING:
Plan to Share IPD: No